CLINICAL TRIAL: NCT02949271
Title: Comparison of Programmed Intermittent Epidural Boluses With Continuous Epidural Infusion for Maintenance of Labor Analgesia
Brief Title: Comparison of PIEB vs CEI for Labor Analgesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: Pro00077123
Record Dates: First submitted 2016-10-25; First posted 2016-10-31 (Estimated); Results first posted 2019-01-11 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Labor Pain
Keywords: epidural analgesia
MeSH Terms: conditions — Labor Pain | interventions — Ropivacaine; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Programmed Intermittent Epidural Bolus (Active Comparator): Epidural catheters will be placed at the L3/4 or L4/5 interspace with 4 cm of catheter being left in the epidural space. Epidural analgesia will be initiated and maintained with a solution of ropivacaine 0.1% with fentanyl 2 mcg/ml. After the initial epidural loading dose of 20 mL is administered in incremental fashion, patients will receive either 6 mL every 45 minutes in the PIEB arm (first bolus 30 minutes after epidural initiation). All study participants will be provided with PCEA set to 8mL boluses with a 10-minute lockout period. The maximum amount of PCEA analgesia will be set to a 1-hour maximum of 45mL.
  Interventions: Other: Programmed Intermittent Epidural Bolus; Drug: Ropivacaine; Drug: Fentanyl
- Continuous Epidural Infusion (Active Comparator): Epidural catheters will be placed at the L3/4 or L4/5 interspace with 4 cm of catheter being left in the epidural space. Epidural analgesia will be initiated and maintained with a solution of ropivacaine 0.1% with fentanyl 2 mcg/ml. After the initial epidural loading dose of 20 mL is administered in incremental fashion, patients will receive 8mL/hr of continuous infusion beginning immediately after the loading dose for the maintenance of analgesia in the CEI arm. All study participants will be provided with PCEA set to 8mL boluses with a10-minute lockout period. The maximum amount of PCEA analgesia will be set to a 1-hour maximum of 45mL.
  Interventions: Other: Continuous Epidural Infusion; Drug: Ropivacaine; Drug: Fentanyl

INTERVENTIONS:
Other: Programmed Intermittent Epidural Bolus
  Arms: Programmed Intermittent Epidural Bolus
Other: Continuous Epidural Infusion
  Arms: Continuous Epidural Infusion
Drug: Ropivacaine
Drug: Fentanyl

SUMMARY:
The aim of this prospective, doubled-blinded randomized study is to compare two modes of epidural analgesia delivery, programmed intermittent epidural boluses (PIEB) versus continuous epidural infusion (CEI) with patient controlled epidural analgesia (PCEA) dosing, for providing labor epidural analgesia. The primary outcome will be the volume of local anesthetic received through PCEA. Secondary outcomes will measure time to first PCEA bolus, labor pain scores, degree of motor blockade, mode of delivery, PCEA attempts and ratio of successful to unsuccessful attempts, frequency of hypotension, duration of first and second stages of labor and level of patient satisfaction. The investigator plans to enroll 120 nulliparous participants at 2-5 com cervical dilation, with 60 patients to each arm. The subject will be assigned to receive either delivery of epidural medication ropivacaine 0.1% with fentanyl 2mcg/mL with PIEB + PCEA dosing method or CEI + PCEA. Continuous data will be analyzed using the Kruskal-Wallis test or t-test as appropriate. Categorical data will be analyzed using Chi-square test or Fisher's exact test as appropriate.

DETAILED DESCRIPTION:
Labor pain during childbirth is regarded as one of the most painful experiences in a woman's life with the potential to cause lasting emotional and psychological effects. Childbirth has also been associated with the development of chronic pain with the prevalence of between 4-10% after cesarean section and 6-18% after vaginal delivery. Hence, effective management of labor pain is instrumental in preventing the development of life altering chronic pain in women of childbearing age. Maintaining epidural analgesia with combined local anesthetic and an opioid is considered extremely safe and leads to superior neonatal and maternal short and long-term outcomes. Historically, maintenance of epidural analgesia involved intermittent provider-administered bolus injections, patient controlled epidural analgesia (PCEA) and continuous epidural infusions (CEI) with or without PCEA for breakthrough pain or discomfort. CEI has been shown to provide consistent analgesia in addition to improved patient satisfaction and reduced workload for the anesthesia providers. However, CEI is associated with greater local anesthetic consumption and increased maternal motor blockade. Increased motor block is associated with reduced mobility, decreased pelvic muscle tone and impaired ability for the parturient to adequately Valsalva during the second stage of labor. Motor blockade is also associated with increased incidence of shoulder dystocia and instrumental deliveries, which precipitate birth trauma to the fetus and the mother. Achieving adequate analgesia during labor, without compromising motor function is critical for optimizing both short-term and long-term outcomes for the mother and the neonate.

A more novel approach to labor analgesia involves the administration of small, programmed intermittent epidural boluses (PIEB) with PCEA dosing for breakthrough pain. Preliminary studies have indicated that PIEB could be a superior method of labor analgesia compared to current standard of care, CEI. A randomized double-blind study by Wong et al. compared CEI and PIEB incorporating the use of PCEA for breakthrough pain in healthy parturients with singleton pregnancies. Results suggested that the cohort receiving PIEB required less local anesthetic use, had similar analgesia and improved patient satisfaction when compared with CEI. Additionally, a subsequent study by Wong et al found that in healthy, term, nulliparous women in spontaneous labor, extending the PIEB interval and increasing volume decreased local anesthetic consumption, PCEA requests or rescue analgesia requirements without increasing patient discomfort or compromising satisfaction. Two subsequent studies allocating women to receive either PIEB or CEI in nulliparous parturients and women terminating pregnancy suggested PIEB recipients experienced less motor blockade when compared to those receiving CEI.

The investigator has recently performed a systematic review and meta-analysis of studies comparing the effects of labor analgesia with either PIEB or CEI with or without PCEA in laboring women. The meta-analysis included 9 studies and evaluated various primary outcomes including: patient satisfaction, required manual anesthesia interventions, labor progression and mode of delivery (vaginal, instrumental or cesarean delivery). Secondary outcomes included: degree of motor blockade, degree of sensory blockade, time to first anesthetic intervention, local anesthetic dose delivered per hour, pruritus, shivering, maternal fever, nausea and vomiting, neonatal Apgar scores at 1 minute and 5 minutes, and umbilical artery and vein pH. PIEB dosing of local anesthetic was associated with reduced local anesthetic consumption, decreased required anesthetic interventions, and an improvement in maternal satisfaction in comparison to laboring women receiving CEI. Pooled results indicated that PIEB and CEI were comparable with regard to the duration of first stage labor, but there was a statistically significant 22 min reduction in the length of stage two of labor with PIEB. Similarly, this review did not suggest statistically significant differences in cesarean delivery rate or required anesthetic intervention between CEI and PIEB. There were several limitations to these preliminarily studies. While, each of the 9 studies reported at least one primary outcome listed in the systematic review, none of the studies included all primary outcomes. Additionally, most studies only involved nulliparous women, which may limit the ability to apply results to multiparous women. Furthermore, many of these studies involved the use of two pumps, one to deliver CEI or PEIB and another to deliver PCEA in a research setting, or involved the use of non-commercially available research pumps.

Currently the CADD solis v 3.0 pump system has been upgraded to allow the co-administration of epidural anesthesia with PIEB or CEI and PCEA. This new technology has been available on the labor and delivery unit of Duke University Medical Center as the standard of care since March 2015. This new pump differs from those used in the preliminary studies, which utilized a two-pump approach to administer PIEB or CEI and PCEA for labor pain relief. Preliminary studies have not identified optimal PIEB settings, bolus volumes, lock out intervals, or drug concentrations, which represents a gap in literature at the present time. The investigator performed a retrospective study to explore whether PIEB was associated with reduced LA use, PCEA use and rescue analgesia in comparison to CEI in laboring women. The investigator also assessed whether PIEB decreased the number of instrumental deliveries and reduced motor blockade, which serves as an impediment to the progression of labor. The study divided patients into three groups. The first received CEI 5mL/hour, the second received PIEB 5mL every 60 min, the third used PIEB of 3mL every 30 min. Each group had access to PCEA set to 5 mL boluses with an 8-minute lockout period and maximum of 35mL per hour. The results of the study did not suggest what was expected as the study revealed no statistically significant difference between the LA consumption, amount of motor blockade or mode of delivery for patients receiving CEI or PEIB when using the single pump system instead of two-pump system employed by prior studies. However, this study did suggest patients who received PIEB regimen of 3mL every 30 minutes used a lower PCEA volume than patients receiving CEI. Patients receiving PEIB regimens had more attempts/PCEA given than the CEI patients and the PIEB 3ml/30 minute group had more unsuccessful PCEA attempts/hour than CEI recipients.

This study, unlike prior studies comparing PIEB vs. CEI with PCEA, used more concentrated solutions consisting of double the concentration and half the volume of bupivacaine. One of the investigators speculations is that larger boluses of a more dilute LA may have improved dissemination in the epidural space and thus improved analgesia. This study interpreted PCEA attempts/given and the number of unsuccessful PCEA attempts/hour as reflections of patient pain or discomfort, as an attempt is interpreted as an effort to achieve better pain relief. Another way to interpret the aforementioned PCEA attempts is as representation of the amount of time a patient "locked out" or prevented from receiving additional boluses of PCEA. Hence, a limitation of this study is the fact that patient satisfaction scores were not collected as they could help distinguish whether attempts reflect the lockout period or inadequate analgesia. Other limitations of this retrospective study include the fact that explicit instructions about how to properly use the PCEA was not standardized, and the fact that patient satisfaction or pain scores were not garnered due to the study's retrospective nature. Probably one of the most significant limitations of this study was the fact that patients were not randomized to treatment groups. Hence, the providers chose the analgesia received. On the other hand, another retrospective study utilizing a more dilute concentration of local anesthetic reported reduced need for physician interventions with PIEB compared to CEI. The investigators have recently switched the local anesthetic in our practice from bupivacaine 0.125 % to a more dilute concentration of ropivacaine 0.1% mixed with fentanyl 2 mcg/ml. The investigator therefore aims to prospectively study if the use of PIEB with the new epidural solution would be associated with improved analgesia compared to a regimen using CEI.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology (ASA) class 2 and 3 women
* Nulliparous
* Age > 18 yrs
* gestational age > 36 weeks
* singleton pregnancies
* vertex pregnancies
* spontaneous labor or scheduled induction of labor
* cervical dilatation 2-5 cm at time of epidural placement
* Pain score > 5

Exclusion Criteria:

* BMI > 50 kg/m2
* history of past or current intravenous drug or chronic opioid abuse
* chronic analgesic use
* allergy or contraindication to any study medications
* any maternal or fetal condition requiring planned assisted stage 2 delivery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2016-11-08 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf S Habib, MBBCh, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vermelis JM, Wassen MM, Fiddelers AA, Nijhuis JG, Marcus MA. Prevalence and predictors of chronic pain after labor and delivery. Curr Opin Anaesthesiol. 2010 Jun;23(3):295-9. doi: 10.1097/aco.0b013e32833853e8. PMID 20446346
- [Background] Leighton BL, Halpern SH. The effects of epidural analgesia on labor, maternal, and neonatal outcomes: a systematic review. Am J Obstet Gynecol. 2002 May;186(5 Suppl Nature):S69-77. doi: 10.1067/mob.2002.121813. PMID 12011873
- [Background] Wong CA, Scavone BM, Peaceman AM, McCarthy RJ, Sullivan JT, Diaz NT, Yaghmour E, Marcus RJ, Sherwani SS, Sproviero MT, Yilmaz M, Patel R, Robles C, Grouper S. The risk of cesarean delivery with neuraxial analgesia given early versus late in labor. N Engl J Med. 2005 Feb 17;352(7):655-65. doi: 10.1056/NEJMoa042573. PMID 15716559
- [Background] Thornton JG, Capogna G. Reducing likelihood of instrumental delivery with epidural anaesthesia. Lancet. 2001 Jul 7;358(9275):2. doi: 10.1016/s0140-6736(00)05295-8. No abstract available. PMID 11454363
- [Background] Wong CA, McCarthy RJ, Hewlett B. The effect of manipulation of the programmed intermittent bolus time interval and injection volume on total drug use for labor epidural analgesia: a randomized controlled trial. Anesth Analg. 2011 Apr;112(4):904-11. doi: 10.1213/ANE.0b013e31820e7c2f. PMID 21430035
- [Background] Capogna G, Camorcia M, Stirparo S, Farcomeni A. Programmed intermittent epidural bolus versus continuous epidural infusion for labor analgesia: the effects on maternal motor function and labor outcome. A randomized double-blind study in nulliparous women. Anesth Analg. 2011 Oct;113(4):826-31. doi: 10.1213/ANE.0b013e31822827b8. Epub 2011 Jul 25. PMID 21788309
- [Background] Leone Roberti Maggiore U, Silanos R, Carlevaro S, Gratarola A, Venturini PL, Ferrero S, Pelosi P. Programmed intermittent epidural bolus versus continuous epidural infusion for pain relief during termination of pregnancy: a prospective, double-blind, randomized trial. Int J Obstet Anesth. 2016 Feb;25:37-44. doi: 10.1016/j.ijoa.2015.08.014. Epub 2015 Oct 1. PMID 26431778
- [Background] George RB, Allen TK, Habib AS. Intermittent epidural bolus compared with continuous epidural infusions for labor analgesia: a systematic review and meta-analysis. Anesth Analg. 2013 Jan;116(1):133-44. doi: 10.1213/ANE.0b013e3182713b26. Epub 2012 Dec 7. PMID 23223119
- [Background] Tien M, Allen TK, Mauritz A, Habib AS. A retrospective comparison of programmed intermittent epidural bolus with continuous epidural infusion for maintenance of labor analgesia. Curr Med Res Opin. 2016 Aug;32(8):1435-40. doi: 10.1080/03007995.2016.1181619. Epub 2016 May 20. PMID 27100210
- [Background] McKenzie CP, Cobb B, Riley ET, Carvalho B. Programmed intermittent epidural boluses for maintenance of labor analgesia: an impact study. Int J Obstet Anesth. 2016 May;26:32-8. doi: 10.1016/j.ijoa.2015.11.005. Epub 2015 Nov 27. PMID 26775896

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study took place at Duke University Medical Center from November 2016-November 2017.
Pre-assignment Details: 298 were assessed for eligibility and 119 subjects were excluded due to not meeting exclusion criteria.
Groups:
- Programmed Intermittent Epidural Bolus: Epidural catheters will be placed at the L3/4 or L4/5 interspace with 4 cm of catheter being left in the epidural space. Epidural analgesia will be initiated and maintained with a solution of ropivacaine 0.1% with fentanyl 2 mcg/ml. After the initial epidural loading dose of 20 mL is administered in incremental fashion, patients will receive either 6 mL every 45 minutes in the PIEB arm (first bolus 30 minutes after epidural initiation). All study participants will be provided with PCEA set to 8mL boluses with a 10-minute lockout period. The maximum amount of PCEA analgesia will be set to a 1-hour maximum of 45mL.
  Programmed Intermittent Epidural Bolus
  Ropivacaine
  Fentanyl
- Continuous Epidural Infusion: Epidural catheters will be placed at the L3/4 or L4/5 interspace with 4 cm of catheter being left in the epidural space. Epidural analgesia will be initiated and maintained with a solution of ropivacaine 0.1% with fentanyl 2 mcg/ml. After the initial epidural loading dose of 20 mL is administered in incremental fashion, patients will receive 8mL/hr of continuous infusion beginning immediately after the loading dose for the maintenance of analgesia in the CEI arm. All study participants will be provided with PCEA set to 8mL boluses with a10-minute lockout period. The maximum amount of PCEA analgesia will be set to a 1-hour maximum of 45mL.
  Continuous Epidural Infusion
  Ropivacaine
  Fentanyl
Period: Overall Study
Arm/Group | Programmed Intermittent Epidural Bolus | Continuous Epidural Infusion
Started | 90 | 89
Completed | 61 | 59
Not Completed | 29 | 30
Not completed — Lack of Efficacy | 5 | 4
Not completed — Lost to Follow-up | 3 | 6
Not completed — Physician Decision | 5 | 5
Not completed — Protocol Violation | 6 | 3
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Delivered prior to intervention | 7 | 9
Not completed — Outside the window for cervical dilation | 2 | 3

BASELINE CHARACTERISTICS:
Population: Participants who completed the study
Groups:
- Total: Total of all reporting groups
Arm/Group | Programmed Intermittent Epidural Bolus | Continuous Epidural Infusion | Total
Number analyzed (Participants) | 61 | 59 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.5 (5.0) | 29.8 (5.3) | 29.2 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 59 | 120
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 5
  Not Hispanic or Latino | 60 | 55 | 115
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 1 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 20 | 38
  White | 37 | 38 | 75
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 61 | 59 | 120

OUTCOME MEASURES:

1. Primary Outcome: Volume of Local Anesthetic Received Through Patient Controlled Epidural Analgesia (PCEA) Per Hour
Description: The volume of local anesthetic that the patient received through activation of the patient-controlled epidural analgesia system per hour.
Time Frame: duration of labor, up to 24hrs
Measure: Median (Inter-Quartile Range); unit: milliliters per hour
Arm/Group | Programmed Intermittent Epidural Bolus | Continuous Epidural Infusion
Number analyzed (Participants) | 61 | 59
milliliters per hour | 4.03 [2.15 to 7.07] | 4.52 [2.99 to 8.63]
Statistical Analysis 1: Comparison: Programmed Intermittent Epidural Bolus vs Continuous Epidural Infusion; Test type: Other; p = 0.17, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Volume of Local Anesthetic Required Per Hour
Description: The total volume of local anesthetic that the patient received from the CAPP pump per hour.
Time Frame: duration of labor, up to 24hrs
Measure: Median (Inter-Quartile Range); unit: milliliters per hour
Arm/Group | Programmed Intermittent Epidural Bolus | Continuous Epidural Infusion
Number analyzed (Participants) | 61 | 59
milliliters per hour | 11.49 [9.21 to 14.84] | 12.38 [10.45 to 17.03]
Statistical Analysis 1: Comparison: Programmed Intermittent Epidural Bolus vs Continuous Epidural Infusion; Test type: Other; p = 0.18, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Time to First Patient Controlled Epidural Analgesia (PCEA) Bolus
Time Frame: duration of labor, up to 24hrs
Population: Data not collected since it required extracting data that are not collected as part of standard practice and study team was not available sometimes when the patient delivered and this data had to be collected then before the pump was used for another patient.
Arm/Group | Programmed Intermittent Epidural Bolus | Continuous Epidural Infusion
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Maximum Reported Labor Pain Score
Description: Measured using a verbal analog pain scale of 1-10, where 0=no pain and 10=worst possible pain.
Time Frame: duration of labor, up to 24hrs
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Programmed Intermittent Epidural Bolus | Continuous Epidural Infusion
Number analyzed (Participants) | 61 | 59
score on a scale | 3 [0 to 6] | 2 [0 to 4]
Statistical Analysis 1: Comparison: Programmed Intermittent Epidural Bolus vs Continuous Epidural Infusion; Test type: Other; p = 0.27, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Degree of Motor Blockade Measured as Lowest Recorded Modified Bromage Score
Description: The Modified Bromage Score ranges from 1-5. 1 = complete block, 2 = almost complete block, 3 = partial block, 4 = detectable weakness of hip flexion, and 5 = no detectable weakness of hip flexion while supine.
Time Frame: duration of labor, up to 24hrs
Population: Data not collected on 10 participants in the Programmed Intermittent Epidural Bolus group and in 7 in the continuous epidural infusion group.
Measure: Count of Participants; unit: Participants
Arm/Group | Programmed Intermittent Epidural Bolus | Continuous Epidural Infusion
Number analyzed (Participants) | 51 | 52
Participants
  Score of 5 | 37 | 26
  Score of 4 | 9 | 20
  Score of 3 | 4 | 3
  Score of 2 | 1 | 2
  Score of 1 | 0 | 1
Statistical Analysis 1: Comparison: Programmed Intermittent Epidural Bolus vs Continuous Epidural Infusion; Test type: Other; p = 0.28, Chi-squared

6. Secondary Outcome: Total Number of Subjects Experiencing Each Mode of Delivery
Description: Modes of delivery: spontaneous vaginal delivery (SVD), assisted vaginal delivery (AVD), and caesarean delivery (CD)
Time Frame: duration of labor, up to 24hrs
Measure: Count of Participants; unit: Participants
Arm/Group | Programmed Intermittent Epidural Bolus | Continuous Epidural Infusion
Number analyzed (Participants) | 61 | 59
Participants
  SVD | 41 | 37
  AVD | 5 | 5
  CD | 15 | 17
Statistical Analysis 1: Comparison: Programmed Intermittent Epidural Bolus vs Continuous Epidural Infusion; Test type: Other; p = 0.85, Chi-squared

7. Secondary Outcome: Number of Patient Controlled Epidural Analgesia (PCEA) Attempts
Description: Determined by the number of times subject activates the PCEA pump
Time Frame: duration of labor, up to 24hrs
Measure: Median (Inter-Quartile Range); unit: attempts
Arm/Group | Programmed Intermittent Epidural Bolus | Continuous Epidural Infusion
Number analyzed (Participants) | 61 | 59
attempts | 0.75 [0.33 to 1.84] | 0.63 [0.42 to 1.35]
Statistical Analysis 1: Comparison: Programmed Intermittent Epidural Bolus vs Continuous Epidural Infusion; Test type: Other; p = 0.53, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Ratio of Patient Controlled Epidural Analgesia (PCEA) Successful Attempts to Unsuccessful Attempts
Description: Ratio generated by the number of times subjects activates PCEA and receives additional anesthetic compared with times subject activates PCEA and does not receive additional anesthetic.
Time Frame: duration of labor, up to 24hrs
Measure: Median (Inter-Quartile Range); unit: ratio of attempts
Arm/Group | Programmed Intermittent Epidural Bolus | Continuous Epidural Infusion
Number analyzed (Participants) | 61 | 59
ratio of attempts | 0.17 [0.10 to 0.30] | 0.12 [0.08 to 0.18]
Statistical Analysis 1: Comparison: Programmed Intermittent Epidural Bolus vs Continuous Epidural Infusion; Test type: Other; p = 0.03, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Number of Subjects Experiencing Hypotension Requiring Vasopressor Treatment
Description: Number of patients who needed a vasopressor medication to treat a drop in blood pressure
Time Frame: duration of labor, up to 24 hrs
Measure: Count of Participants; unit: Participants
Arm/Group | Programmed Intermittent Epidural Bolus | Continuous Epidural Infusion
Number analyzed (Participants) | 61 | 59
Participants | 8 | 3
Statistical Analysis 1: Comparison: Programmed Intermittent Epidural Bolus vs Continuous Epidural Infusion; Test type: Other; p = 0.21, Chi-squared

10. Secondary Outcome: Duration of Second Stage of Labor
Time Frame: duration of labor, up to 24hrs
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Programmed Intermittent Epidural Bolus | Continuous Epidural Infusion
Number analyzed (Participants) | 61 | 59
minutes | 44 [15 to 119] | 63 [27 to 130]

11. Secondary Outcome: Number of Subjects Who Were Satisfied With Procedure
Description: Determined using a 5-point scale where 1=very dissatisfied, 2=dissatisfied, 3=neutral, 4=satisfied, 5=very satisfied. Subjects were considered "satisfied" if selected "very satisfied" or "satisfied" on the patient questionnaire.
Time Frame: duration of labor, up to 24hrs
Measure: Count of Participants; unit: Participants
Arm/Group | Programmed Intermittent Epidural Bolus | Continuous Epidural Infusion
Number analyzed (Participants) | 61 | 59
Participants
  Very satisfied | 35 | 39
  Satisfied | 9 | 3
Statistical Analysis 1: Comparison: Programmed Intermittent Epidural Bolus vs Continuous Epidural Infusion; Test type: Other; p = 0.08, Chi-squared

ADVERSE EVENTS:
Time Frame: Duration of labor, up to 24hrs
Arm/Group | Programmed Intermittent Epidural Bolus | Continuous Epidural Infusion
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/59
Other Adverse Events (participants affected / at risk) | 8/61 | 3/59
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Programmed Intermittent Epidural Bolus (N=61) | Continuous Epidural Infusion (N=59)
Hypotension (Cardiac disorders) | 8 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-22): https://cdn.clinicaltrials.gov/large-docs/71/NCT02949271/Prot_SAP_000.pdf